CLINICAL TRIAL: NCT06646172
Title: Liposomal Bupivacaine and Bupivacaine Alone Transverse Thoracic Muscle Plane Blocks in Median Sternotomy: a Prospective, Single-blind, Randomized Controlled Study
Brief Title: Liposomal Bupivacaine and Bupivacaine for TTMPB in Median Sternotomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Tianzhu Liu, Principal Investigator, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Tongji Hospital102114-3
Record Dates: First submitted 2024-10-12; First posted 2024-10-17 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Median Sternotomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mixture of liposome bupivacaine and bupivacaine hydrochloride (Experimental): The same anesthesiologist with experience in regional block was used for ultrasound guided bilateral transverse thoracic muscle plane block (T4-5 interstital space, paracentral transverse axis position). According to the literature, in this study, 1.33% bupivacaine liposome 10 mL + 0.5% bupivacaine hydrochloride 10 ml was used.
  Interventions: Procedure: Transverse thoracic muscle plane block (TTMPB) using liposomal bupivacaine and bupivacaine mixture
- Bupivacaine hydrochloride alone (Active Comparator): The same anesthesiologist with experience in regional block was used for ultrasound guided bilateral transverse thoracic muscle plane block (T4-5 interstital space, paracentral transverse axis position). According to the literature, in this study, 0.5% bupivacaine 20ml was used.
  Interventions: Procedure: Transverse thoracic muscle plane block (TTMPB) using bupivacaine hydrochloride

INTERVENTIONS:
Procedure: Transverse thoracic muscle plane block (TTMPB) using liposomal bupivacaine and bupivacaine mixture — Liposomal bupivacaine and bupivacaine mixture were used for transverse thoracic muscle plane block (TTMPB) in experimental group.
  Arms: Mixture of liposome bupivacaine and bupivacaine hydrochloride
Procedure: Transverse thoracic muscle plane block (TTMPB) using bupivacaine hydrochloride — Bupivacaine hydrochloride was used for transverse thoracic muscle plane block (TTMPB) in active control group.
  Arms: Bupivacaine hydrochloride alone

SUMMARY:
In light of the ongoing controversy surrounding the efficacy of bupivacaine liposomes, our study was designed to investigate, for the first time, the differential postoperative analgesic effects between bupivacaine liposomes combined with bupivacaine hydrochloride and bupivacaine hydrochloride alone in transverse thoracic muscle plane block treatment. The aim is to provide evidence-based medical guidance for drug selection in regional block local anesthesia.

DETAILED DESCRIPTION:
Median thoracic incision is a common method in cardiac surgery for valve replacement, coronary artery bypass and large vessel reconstruction. This kind of surgery is generally more traumatic, with obvious pain stimulation and intense stress response. Compared with other types of surgery, thoracotomy often requires larger doses of opioid analgesics, but excessive use of perioperative opioids has significant adverse effects on postoperative recovery, including sedation, constipation, nausea, addiction and respiratory depression. In addition, improper management of perioperative acute pain during thoracotomy may turn into chronic pain, which will seriously affect patients' postoperative quality of life. For pain management in thoracotomy surgery, the previous practice was to use thoracic epidural continuous catheterization to perform intradural block, but due to the narrow vertebral space in the thoracic vertebrae, this technique is difficult to operate, and for cardiac surgery, individual heparinization requirements of extracorporeal circulation during the operation may greatly increase the possibility of epidural catheter hematoma. Other studies have shown that thoracic epidural block may further lead to sympathetic block, which increases the complexity of perioperative hemodynamic management and concerns the possibility of cerebrovascular accidents.

Transversus Thoracic Plane block (TTP) is a relatively new fascial plane block method. Ultrasound visualization guidance significantly improved the safety of transversus thoracic plane block, and precise injection of local anesthesia drugs could provide perfect analgesia for the anterior branches of the second to sixth intercostal nerves. At the same time, the dosage of other analgesic drugs including opioids can be reduced to reduce the occurrence of related complications [9, 10]. Compared with multimodal analgesia alone, transverse thoracic muscle plane block can significantly reduce postoperative opioid dose. Unlike paravertebral block, the target of the transverse thoracic plane block is the distal branch of the anterior spinal nerve, so there is no risk of sympathetic block, and the injection site is far from the foramen, and there is no risk of intraspinal block or general spinal anesthesia. In view of its high effectiveness and safety, it has been successfully applied in adults and children with median thoracotomy and achieved good perioperative analgesic effects. According to the literature, the transverse thoracic plane block can also be used for the analgesic management of sternal fracture, rib fracture, sternotomy, chronic pain, and the medial incision of breast surgery.

Long-acting amide local anesthetics have been used for surgical incision infiltration anesthesia and shoulder intermuscular groove regional block anesthesia. Although bupivacaine can meet the regional anesthesia requirements for most surgeries, bupivacaine is more likely to cause serious cardiotoxicity when given the same dose as ropivacaine. Bupivacaine and ropivacaine, commonly used local anesthetics for regional block, are similar in terms of sensory action, duration, and blocking effect, but Ropivacaine has greater sensory-motor selectivity, less central nervous system and cardiac toxicity, wider safe dose range, lower reinforcement effect, and longer motor block duration. Therefore, in the current domestic regional block anesthesia technology, the application of both in regional block is more extensive.

Liposomal bupivacaine is a long-acting local anesthetic drug prepared by liposomal technology with slow-release characteristics. It has been reported that the action time of a single administration of bupivacaine liposomal is as high as 72 hours. The drug was approved by the U.S. Food and Drug Administration in October 2011 for postoperative pain management and in April 2018 for nerve block producing regional anesthesia. Compared with bupivacaine, most current research results suggest that the blocking effect of bupivacaine liposomes is not significantly superior to that of standard bupivacaine. However, other studies have suggested that bupivacaine liposomes have a significant advantage in reducing early postoperative opioid use. A non-inferior study of bupivacaine liposome and bupivacaine hydrochloride combined with bupivacaine hydrochloride intermuscular brachial plexus block in patients with total shoulder arthroplasty by Neil A Hanson et al. found that although there was a statistically significant reduction in opioid use on day 3 after surgery, However, the cumulative use of opioids in the bupivacaine hydrochloride group within 3 days after surgery did not show significant inferiority.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-90 years;
* ASA Class I ~ III;
* Patients undergoing elective median sternotomy.

Exclusion Criteria:

* Emergency surgery;
* Re-operation;
* Coagulation dysfunction;
* Preoperative left ventricular function was poor (ejection fraction <35%);
* Systemic infection or injection site infection;
* Neuromuscular diseases;
* Mental illness;
* Dependence on psychotropic drugs;
* Allergic to bupivacaine liposomes and bupivacaine;
* Patients have participated in previous trials or have been determined by a surgeon or anesthesiologist to be unsuitable for randomization;
* Failure to obtain written informed consent from the patient or his/her representative

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2026-10-12 (Estimated)

PRIMARY OUTCOMES:
Third-day opioid consumption | 48-72 hours after surgery
  Opioid consumption was converted to Milligram morphine equivalent (MME) using the analgesic Drug Equivalence calculator.

SECONDARY OUTCOMES:
Cumulative opioid consumption 72 hours after surgery | 0-72 hours after surgery
  Opioid consumption was converted to Milligram morphine equivalent (MME) using the analgesic Drug Equivalence calculator.
Numerical rating scales, NRS | 24 hours, 48 hours and 72 hours after surgery
  Numerical rating scales, NRS: 0-10 A score of 0 is reported as completely painless, and a score of 10 is reported as the most intolerable pain.
Sensory block resolution time | 0-72 hours after surgery
  Time of resolution of numbness in the sternum skin.
Consumption of acetaminophen | 0-72 hours after surgery
  Acetaminophen requirement after surgery.
Consumption of rescue opioid administration | 0-72 hours after surgery
  Rescue opioid is administrated if the NRS > 4
Patient satisfaction | 0-72 hours during and after surgery
  Patient satisfaction with postoperative pain management. (0-5, 0 is very dissatisfied and 5 is very satisfied)
Adverse reactions | 0-72 hours during and after surgery
  Adverse reactions related to block procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Mei Wei, M.D., Study Director — Tongji Hospital
Locations (1):
- Tianzhu Liu, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No